CLINICAL TRIAL: NCT01442727
Title: Selenite in the Detoxification of Arsenic and the Prevention of Arsenical Melanosis and Cancers Amongst Bangladeshi Arsenicosis Patients: A 48-week, Randomized, Double-blinded, Placebo-controlled Phase III Trial
Brief Title: Selenium in the Treatment of Arsenic Toxicity and Cancers
Acronym: SETAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Julian Spallholz, Professor of Nutrition & Biochemistry, Division of Nutritional Sciences, College of Human Sciences, Texas Tech University., Texas Tech University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TTU-JES-1; 1R21CA117111-01 (NIH); ROG-06-098-01 (Other Grant/Funding Number: The American Cancer Society)
Record Dates: First submitted 2011-09-22; First posted 2011-09-28 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Arsenical Melanosis; Arsenical Keratosis; Arsenical Cancers; Arsenicosis; Arsenic Exposure; Arsenic Toxicity; Arsenic Poisoning
Keywords: arsenical melanosis; arsenical melanoses; arsenical keratosis; arsenical keratoses; arsenical cancer; arsenic cancers; arsenic; arsenicosis; arsenic exposure; arsenic toxicity; arsenic poisoning; drinking water; selenium; selenite; sodium selenite
MeSH Terms: conditions — Arsenic Poisoning | interventions — Sodium Selenite; Selenium; Selenious Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients who receive control (placebo)
  Interventions: Drug: placebo
- Selenium (Active Comparator): Patients who receive treatment (selenium)
  Interventions: Drug: sodium selenite

INTERVENTIONS:
Drug: sodium selenite — 200 micrograms (µg) of selenium in the form of sodium selenite; capsule form consumed once daily with breakfast.
  Other Names: selenium; selenite
  Arms: Selenium
Drug: placebo — dicalcium phosphate capsule matching the selenium capsule in appearance; consumed once daily with breakfast
  Arms: Placebo

SUMMARY:
Context: Approximately 100 million people throughout the world consume water contaminated with arsenic at levels above carcinogenic thresholds, including 40 million in Bangladesh alone, with up to one-fourth of deaths attributed to arsenic exposure in the worst-affected regions. There are no proven therapies for treating chronic arsenic toxicity or for preventing arsenical cancers. Selenium has been known to counter arsenic toxicity in a variety of animal models. The investigators have recently shown in animals and humans that this effect is mediated by the formation of [(GS)2AsSe]- , the seleno-bis(S-glutathionyl) arsinium ion, which is then rapidly excreted via the hepatobiliary system. Concurrently, two Phase II studies in China and Bangladesh have suggested clinical benefit to selenium supplementation in arsenicosis patients.

Objective: To assess whether daily selenium supplementation counters arsenic toxicity in patients exposed to drinking water arsenic. If proven effective, selenium supplementation might be safely and cost-effectively implemented in the worst-affected localities.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Bangladesh in an arsenic-affected region (Chandpur)
* Age between 12 and 55
* Exposure to arsenic in home drinking water greater than 50 ug/L.
* Arsenical melanosis on the torso confirmed by epiluminescence microscopy

Exclusion Criteria:

* Recent history or plans to consume selenium-containing supplements
* Anticipated change in home drinking water supply during study period

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 819 (Actual)
Dates: Start 2006-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
changes in arsenical melanosis | 0 weeks (baseline), 24 weeks, and 48 weeks (end)
  Arsenical melanosis was recorded in 4 quadrants of each patients' torsos using the Dermlite epiluminescence microscopy system. The images were then scored in a blinded, randomized fashion by a dermatologist.

SECONDARY OUTCOMES:
changes in blood arsenic levels | week 0, week 24 and week 48
  The levels of arsenic in patients' blood was measured to determine whether intervention had a differential effect.
changes in urinary arsenic levels | week 0, week 24 and week 48
  The levels of arsenic in patients' urine was measured to determine whether intervention had a differential effect.

CONTACTS AND LOCATIONS:
Overall Officials: Julian E Spallholz, PhD, Principal Investigator — Texas Tech University; Paul F La Porte, PhD, Principal Investigator — Pritzker School of Medicine, The University of Chicago; Selim Ahmed, MBBS, FCPS, Principal Investigator — Institute of Child & Mother Health, Dhaka, Bangladesh
Locations (1):
- SETAC Trial Field Office, Kalibari Town, Chandpur District, Bangladesh